CLINICAL TRIAL: NCT04482686
Title: A Phase I Double-Blind Randomized Placebo-Controlled Trial of Combination Therapy to Treat COVID-19 Infection
Brief Title: Trial of Combination Therapy to Treat COVID-19 Infection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ProgenaBiome (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRG-049
Record Dates: First submitted 2020-07-21; First posted 2020-07-22 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: COVID; Covid-19; Corona Virus Infection; Coronavirus Infection; Coronavirus-19; SARS-CoV2; SARS-CoV Infection
MeSH Terms: conditions — COVID-19; Coronavirus Infections; Severe Acute Respiratory Syndrome | interventions — Ivermectin; Doxycycline; Zinc; Zinc Sulfate; Cholecalciferol; Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active Arm (Experimental): Patients will be treated with a combination of Ivermectin, Doxycycline, Zinc, Vitamin D3 and Vitamin C
  Interventions: Drug: Ivermectin; Drug: Doxycycline Hcl; Dietary Supplement: Zinc; Dietary Supplement: Vitamin D3; Dietary Supplement: Vitamin C
- Placebo (Placebo Comparator): Placebo and Vitamin D3, Vitamin C, and Zinc
  Interventions: Dietary Supplement: Zinc; Dietary Supplement: Vitamin D3; Dietary Supplement: Vitamin C

INTERVENTIONS:
Drug: Ivermectin — Treatment days 1, 4, and 8
  Other Names: Soolantra, Stromectol, Sklice
  Arms: Active Arm
Drug: Doxycycline Hcl — 10 day treatment
  Other Names: Doxy-100, Monodox, Oracea, Targadox, Acticlate, Morgidox, Avidoxy, Doryx MPC, Mondoxyne NL, Dory
  Arms: Active Arm
Dietary Supplement: Zinc — 10 Day treatment
  Other Names: Zinc sulphate
Dietary Supplement: Vitamin D3 — 10 day treatment
  Other Names: cholecalciferol-D3
Dietary Supplement: Vitamin C — 10 day treatment
  Other Names: L-ascorbic acid

SUMMARY:
In this trial patients will be treated with either a combination of therapies to treat COVID-19 or a placebo. Treatment will last 10 days, and patients will be followed for 6 months.

DETAILED DESCRIPTION:
Patients in this trial will undergo treatment for 10 days with either a combination of therapies or placebo. They will then be followed for an additional 20 days.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent, demonstrating that the subject understands the procedures required for the study and the purpose of the study
2. Healthy male or female subjects at least 18 years of age
3. Diabetic and obese (BMI > 30) patients will be included in the Trial but randomization will be stratified.
4. Positive test for COVID-19 by RT-PCR or rapid antigen test at screening
5. Subjects must agree to practice at least two highly effective methods of birth control for the duration of the study. One of these must be a barrier method. Exceptions for females and partners of females that are not of childbearing potential. (e.g. surgically sterilized, post-menopausal)
6. Subjects must agree they will attend the treatment facility daily for 10d in the event of failure to attend, the patient will be visited at their home to collect the nasal swab and review data.

Exclusion Criteria:

1. Refusal to sign informed consent form
2. Negative test for COVID-19 by RT-PCR at screening
3. Severe disease symptomatically including pneumonia, respiratory distress, tachypnea, shortness of breath, temperature > 104.0 degrees F, pleuritic pain, or frequent cough.
4. Known drug allergy to any of the investigational medications
5. Currently taking medication with known drug interactions with investigational medications, found in Appendix II
6. Prescription or other antiviral medications
7. Any comorbidities which constitute health risk for the subject including known cardiac arrhythmias - but will be limited to those on hydroxychloroquine
8. Inability to attend daily for 10 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2020-12-09 (Actual); Primary Completion 2022-05-15 (Actual); Study Completion 2022-07-15 (Actual)

PRIMARY OUTCOMES:
Time to Non-Infectivity by RT-PCR | 6 months
  Time to negative RT-PRC result indicating that patient is no longer infective
Time to Symptom progression in days as measured by NEWS scoring system (National Early Warning Score) | 6 months
  Time to reduced symptoms in each treatment group as indicated by NEWS scores, which rate patient status based on a zero to three scale for 8 parameters. These values are added up to create the NEWS score. The lower the NEWS score, the better the patient's clinical condition. Zero is the lowest possible score, whereas 7 or greater represents a high degree of clinical risk.
Time to Symptom improvement as measured by NEWS scoring system (National Early Warning Score) | 6 months
  Time to reduced symptoms in each treatment group as indicated by NEWS scores, which rate patient status based on a zero to three scale for 8 parameters. These values are added up to create the NEWS score. The lower the NEWS score, the better the patient's clinical condition. Zero is the lowest possible score, whereas 7 or greater represents a high degree of clinical risk.
Efficacy of Treatment as measured by Titer | 6 months
  Patients will have serum stored for titer testing to compare antibody levels over time
Efficacy of Treatment as measured by RT-PCR | 10 days
  Number of patients testing negative for SARS-CoV-2 by RT-PCR after 10 days of treatment

SECONDARY OUTCOMES:
Safety of Treatment as Measured by D-Dimer | 6 Months
  Blood D-Dimer levels
Safety of Treatment as Measured by Pro-Calcitonin | 6 Months
  Blood Pro-Calcitonin levels
Safety of Treatment as Measured by C-Reactive Protein | 6 Months
  Blood CRP levels
Safety of Treatment as Measured by Ferritin | 6 Months
  Blood ferritin levels
Safety of Treatment as Measured by Liver Enzymes | 6 Months
  Blood enzyme levels
Safety of Treatment as Measured by Complete Blood Count | 6 Months
  CBC
Safety of Treatment as Measured by Electrolyte Levels | 6 Months
  Blood electrolytes
Safety of Treatment as Measured by Treatment Related Adverse Events | 6 months
  Presence or absence of Grade 3 or high treatment related adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Hazan, MD, Study Director — ProgenaBiome; Thomas Borody, MD, Study Director — Topelia Therpeutics
Locations (1):
- ProgenaBiome, Ventura, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hazan S, Vidal AC, Hulscher N, Goudzwaard A, McCullough PA, Steinberg AA. Cardiac findings in a phase II double-blind randomized placebo-controlled trial of combination therapy (HAZDPac) to treat COVID-19 patients. BMC Cardiovasc Disord. 2024 Dec 19;24(1):710. doi: 10.1186/s12872-024-04376-y. PMID 39702045
- [Derived] Hazan S, Dave S, Gunaratne AW, Dolai S, Clancy RL, McCullough PA, Borody TJ. Effectiveness of ivermectin-based multidrug therapy in severely hypoxic, ambulatory COVID-19 patients. Future Microbiol. 2022 Mar;17:339-350. doi: 10.2217/fmb-2022-0014. Epub 2022 Feb 9. PMID 35135310